CLINICAL TRIAL: NCT02433171
Title: Studies of Methionine-PET and PBR28-PET in Brain Metastases to Differentiate Tumor Recurrence and Radiation Necrosis Following Stereotactic Radiosurgery
Brief Title: Methionine and PBR28-PET (Peripheral Benzodiazepine Receptors) in Brain Metastases Following Radiosurgery
Status: Terminated | Type: Observational
Why Stopped: Lack of available funding.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1401013294
Record Dates: First submitted 2014-12-19; First posted 2015-05-04 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Brain Metastasis
Keywords: regrowth; radiosurgery; radiation necrosis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Melanoma Brain Metastases: Stage 4 cancer patient population with melanoma with brain metastases previously treated with SRS
  Interventions: Procedure: Standard of Care FDG-PET Imaging
- Lung Cancer Brain Metastases: Stage 4 cancer patient population with non-small cell lung cancer with brain metastases previously treated with SRS
  Interventions: Procedure: Standard of Care FDG-PET Imaging

INTERVENTIONS:
Procedure: Standard of Care FDG-PET Imaging — [11C]Methionine [11]. This natural amino acid, and its various fluorinated derivatives, has been widely used in brain tumor studies due to a) high tumor-to-normal brain contrast, and b) its sensitivity to biological functions including amino acid transport and utilization. [11C]PBR28 [12]. This ligand is one of a series of second-generation tracers that bind to TSPO (translocator protein), a protein that is upregulated in activated microglia.
  Other Names: DWI, MRPerfusion, MRSpectroscopy and FDG-PET

SUMMARY:
The goal of this protocol is to evaluate the potential of PET imaging of amino acid transport and microglial activation to improve the differentiation of tumor recurrence and radiation necrosis in patients with brain metastases after treatment with stereotactic radiosurgery (SRS) who have re-growing lesions. These state-of-the-art imaging tools will be used in combination with standard magnetic resonance imaging (MRI), MR spectroscopy (MRS) and FDG-PET (fluorodeoxyglucose).

DETAILED DESCRIPTION:
The investigators hypothesize that by using two different PET tracers, one sensitive to tumor metabolic activity, and one sensitive to inflammatory processes, investigators can separately identify metabolically active tumor from radiation necrosis related inflammation. This can be accomplished with quantitative assessments of tracer uptake using kinetic modeling techniques, as well as by high-resolution imaging to assess the distribution of tracer uptake in the tumor region. All participants in the study will have the receive the same diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with brain metastases from melanoma or non-small cell lung cancer
* Patients must have had SRS and regrowth in at least one lesion > 0.5 cm in greatest dimension and fall into one of two categories: a) patient is deemed clinically appropriate for surgical intervention (biopsy or craniotomy) OR b) patient is asymptomatic and has a life expectancy of > 6 months so that serial follow-up imaging is appropriate
* Willingness to participate in imaging studies
* Able to give informed consent

Exclusion Criteria:

* Subjects with history of prior radiation exposure for research purposes within the past year, such that participation in this study would place them over the FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
* Subjects who are pregnant or currently breastfeeding
* Women of child-bearing age who are sexually active, unless they agree to two forms of contraception, and have a negative urine pregnancy test at screening and on the days of the PET imaging
* Patients unable to undergo MRI with gadolinium-based contrast for standard clinical reasons which include:
* Cardiac pacemaker, aneurysm clip, cochlear implants, Intra Uterine Device (IUD), shrapnel, neurostimulators, defibrillator, artificial heart valve, or history of metal fragments in eyes.
* Pregnancy
* Body size too large for closed MRI
* Known hepatic fibrosis.
* Claustrophobia
* Contraindication to MR contrast agents: eGFR (epidermal growth factor receptor) < 30 by the Cockcroft- Gault formula if > 60 years old or with chronic renal disease
* Anaphylactic allergy to gadolinium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received SRS for melanoma or NSCLC brain metastases with regrowing lesions who are candidates for surgical intervention (biopsy or excision) at the Smilow Cancer Center or are candidates for monitoring by serial imaging will be screened for eligibility and offered enrollment
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Regrowing Tumor Rate from Radiation Effect | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Chiang, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Tran TT, Gallezot JD, Jilaveanu LB, Zito C, Turcu G, Lim K, Nabulsi N, Huang H, Huttner A, Kluger HM, Chiang VL, Carson R. [11C]Methionine and [11C]PBR28 as PET Imaging Tracers to Differentiate Metastatic Tumor Recurrence or Radiation Necrosis. Mol Imaging. 2020 Jan-Dec;19:1536012120968669. doi: 10.1177/1536012120968669. PMID 33147119